CLINICAL TRIAL: NCT03531112
Title: Reducing Binge Eating to Prevent Weight Gain in Black Women: A Pilot Study
Brief Title: Reducing Binge Eating to Prevent Weight Gain in Black Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to COVID-19
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0784; P30DK056350 (NIH)
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-07

CONDITIONS: Binge Eating; Weight Loss; Weight Gain Prevention
MeSH Terms: conditions — Bulimia; Weight Loss

STUDY DESIGN:
Intervention Model Description: The proposed study will use a randomized clinical trial design. A sample of 40 black women who report at least weekly binge eating episodes will be randomized to 2 arms of a 6-month AAT intervention: AAT or a wait-list control group (delayed intervention group). AAT participants will receive an 8-week AAT program using a group format, and will be provided a smart scale (with bluetooth-connection for automatic data reporting) and instructions to weigh themselves daily. Participants will also be provided with weekly tailored feedback on self-weighing frequency and weight change. Assessments will be conducted at 0, 2, and 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appetite Awareness Treatment (AAT) + Lifestyle Modification (LM) (Experimental): Participants will receive an 8-week Appetite Awareness Training (AAT) program using a group format, will be provided a smart scale (with bluetooth connection) and instructions to weigh themselves daily. Participants will also be provided with weekly tailored feedback on self-weighing frequency and weight change. Assessment will be conducted at 0, 2, and 6 months.
  Interventions: Behavioral: Appetite Awareness Treatment + Lifestyle Modification
- Control (No Intervention): Control group participants will receive no intervention in months 1-6, but will be offered the chance to receive an abbreviated form of AAT (4 weeks) following the 6-month assessment.

INTERVENTIONS:
Behavioral: Appetite Awareness Treatment + Lifestyle Modification — The AAT + LM intervention includes 16 60-90 minute group sessions to enable participants to be able to relearn their stomach's hunger signals and begin to obey and monitor functions of satiety. All sessions involve didactic training, review of self-monitoring of eating episodes, interactive activities, and homework assignments to enable participants to practice learned skills. Participants will be provided a workbook, which will include session content, and self-monitoring forms.
  Arms: Appetite Awareness Treatment (AAT) + Lifestyle Modification (LM)

SUMMARY:
The purpose of the proposed study is to pilot a 6-month, cognitive-behavioral binge eating intervention, Appetite Awareness Training (AAT) to reduce binge eating and prevent weight gain for Black women with a BMI > 25 kg/m^2 and with weekly binge eating episodes. Intervention participants will receive a 8-week group AAT intervention, and will also receive bluetooth-connected scales for daily weighing. Participants will also receive tailored feedback on self-weighing frequency and weight change. The investigators will follow-up with participants at six months.

DETAILED DESCRIPTION:
Aim 1. Using an experimental design, examine the feasibility and acceptability of 6-month AAT (N=40) in North Carolina. Forty overweight and obese (BMI ≥ 25 kg/m^2) community-based Black women will be randomized to the AAT intervention or wait-list control (who will eventually receive the intervention). AAT participants will meet weekly for 8 weeks, followed by a 4-month period of daily weighing and weekly tailored feedback only. The study will examine the following: recruitment feasibility, attendance/retention, adherence, satisfaction, and barriers to completion.

Aim 2: At 4 and 6 months, compare changes in (a) binge eating, eating self-efficacy, and depressive symptoms and (b) weight, blood pressure, and waist circumference for participants in the intervention vs. control group.

H_1: Participants in the AAT intervention will report less binge and overeating and gain less weight than those in the control group at 2 and 6 months.

Secondary aim: Examine characteristics (e.g., baseline BMI, severity of binge eating, frequency of self-weighing) related to change in binge eating and weight.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible if they are:

* non-Latino Black women,
* over 18 years of age,
* have a BMI ≥ 25kg/m^2,
* use a Bluetooth-enabled smartphone,
* report at least one binge eating episode weekly, and
* complete the screening.

Exclusion Criteria:

Individuals will be excluded if they:

* are currently pregnant,
* are in substance abuse treatment,
* are involved in another weight reduction program,
* have a history of anorexia,
* are purging,
* are currently in treatment for eating difficulties,
* are concurrent intravenous drug users or consume >4 alcoholic beverages/day.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identify as a female
Enrollment: 20 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Goode, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study terminated prior to enrollment of control participants.
Groups:
- Appetite Awareness Treatment + Lifestyle Modification: Appetite Awareness Treatment (AAT) + Lifestyle Modification (LM): The AAT + LM intervention includes 16 60-90 minute group sessions to enable participants to be able to relearn their stomach's hunger signals and begin to obey and monitor functions of satiety. All sessions involve didactic training, review of self-monitoring of eating episodes, interactive activities, and homework assignments to enable participants to practice learned skills. Participants will be provided a workbook, which will include session content, and self-monitoring forms.
Period: Overall Study
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Started | 20 | 0
Month 4 | 17 | 0
Month 6 (Follow-Up) | 13 | 0
Completed | 13 | 0
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated prior to enrollment of control participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control | Total
Number analyzed (Participants) | 20 | 0 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.8) |  | 46.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 |  | 20
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 20 |  | 20
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 20 |  | 20
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (Recruitment): Total Number of Participants Who Were Eligible and Enrolled in the Study
Description: Recruitment is defined as the number of potential participants screened for study eligibility versus the number of persons who enrolled in the study.
Time Frame: Month 6
Population: Study terminated prior to enrollment of control participants. The number of potential participants screened for study eligibility
Measure: Count of Participants; unit: Participants
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 30 | 0
Participants | 20 |

2. Primary Outcome: Feasibility (Retention): Percentage of Participants Retained in the Study
Description: Percentage of participants retained in the study following enrollment through month 6
Time Frame: Month 6
Population: Study terminated prior to enrollment of control participants.
Measure: Number; unit: percentage of participants
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 20 | 0
percentage of participants | 85 |

3. Primary Outcome: Feasibility (Attendance): Percentage of Sessions That Were Attended
Description: Each session attended by participants was captured. The number of sessions attended for each participant were summed and then divided by the number of total participants and multiplied by 100.
Time Frame: Month 2
Population: Study terminated prior to enrollment of control participants. Data not included for three participants who discontinued.
Measure: Number; unit: percentage of sessions per participant
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 17 | 0
percentage of sessions per participant | 56 |

4. Secondary Outcome: Median Weight Change From Baseline to Month 4
Description: Measured in Kg
Time Frame: Baseline, Month 4
Population: Study terminated prior to enrollment of control participants. Data not included for three participants who discontinued.
Measure: Median (Inter-Quartile Range); unit: Kg
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 17 | 0
Kg | 0 [-1.1 to 1.4] |

5. Secondary Outcome: Median Weight Change From Baseline to Month 6
Description: Measured in Kg
Time Frame: Baseline, Month 6
Population: Study terminated prior to enrollment of control participants. Data not included for seven participants who discontinued.
Measure: Median (Inter-Quartile Range); unit: Kg
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 13 | 0
Kg | -0.2 [-0.9 to 0.5] |

6. Secondary Outcome: Mean Change in Binge Eating Scale Score From Baseline to Month 2
Description: This measure contains 16 questions that describe both behavioral and emotional manifestations of a binge episode. This scale was specifically developed to assess binge eating severity and associated emotional distress in individuals with overweight and obesity. The total score for the measure ranges from 0-46 points with higher scores indicating greater problems with binge eating and lower scores indicating better outcome.
Time Frame: Baseline, Month 2
Population: Data were not collected using the Binge Eating Scale and were instead collected using the Eating Disorder Examination
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Change in Binge Eating Scale Score From Baseline to Month 6
Description: This measure contains 16 questions that describe both behavioral and emotional manifestations of a binge episode. This scale was specifically developed to assess binge eating severity and associated emotional distress in overweight and obese individuals. The total score for the measure ranges from 0-46 points with higher scores indicating greater problems with binge eating and lower scores indicating better outcome.
Time Frame: Baseline, Month 6
Population: Data were not collected using the Binge Eating Scale and were instead collected using the Eating Disorder Examination
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Objective Binge Eating Episodes
Description: Participants were administered the interviewer-based overeating section of the Eating Disorder Examination (EDE) to assess objective binge eating episodes (OBE) (i.e., consumption of an objectively large amount of food and loss of control over eating) within the 28 days prior. Assessed at Baseline, Month 4, and Month 6.
Time Frame: up to 6 months
Population: Study terminated prior to enrollment of control participants.
Measure: Mean (Standard Deviation); unit: binge eating episodes
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
Number analyzed (Participants) | 17 | 0
binge eating episodes
  Baseline | 6.5 (7.8) |
  Month 4 | 2.1 (5.1) |
  Month 6 | 2.6 (6.9) |

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent through Visit 3, an approximate total of up to 6 months.
Description: Study terminated prior to enrollment of control participants.
Arm/Group | Appetite Awareness Treatment + Lifestyle Modification | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/20 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03531112/Prot_SAP_000.pdf